CLINICAL TRIAL: NCT05081583
Title: Clinical Evaluation of the Pharmacokinetic Goldenseal-Metformin Interaction in Diabetic Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18889-002; U54AT008909 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Interaction, Adverse Herb-Drug; Diabetes Mellitus, Type 2
Keywords: pharmacokinetics; natural product-drug interactions; transporters
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study Arm 1: Baseline (Experimental): An anticipated twenty type 2 diabetic subjects (10 males, 10 females) will be administered a single dose of midazolam (0.5 mg) intravenously via a peripherally inserted catheter in conjunction with their daily oral administration of metformin. Plasma and urine will be collected from 0-24 hours post-midazolam administration. Participants will take their metformin as prescribed for the entirety of the study with no interruption in pharmacotherapy.
  Interventions: Drug: Midazolam Hcl 1Mg/Ml Inj
- Study Arm 2: Acute Goldenseal Exposure (Experimental): For Arm 2, the same 20 subjects will be administered a single dose of goldenseal (3.3 g) orally 30 minutes prior to administration of midazolam (as described in Arm 1). Plasma and urine will be collected in a manner identical to that in Arm 1. With respect to midazolam administration, a washout period of 7 days will separate Arm 2 from Arm 1.
  Interventions: Drug: Midazolam Hcl 1Mg/Ml Inj; Dietary Supplement: Goldenseal (Hydrastis canadensis)
- Study Arm 3: Chronic Goldenseal Exposure (Experimental): For Arm 3, the same 20 subjects will be administered goldenseal (1.1 g) orally three times daily for 27 days. On the 28th day, participants will be administered the goldenseal three times daily, as well as the single dose of midazolam (as described in Arm 1). Plasma and urine will be collected in a manner identical to that in Arm 1. A designated washout period for midazolam will not be necessary to separate Arm 3 from Arm 2 since there will be 27 days of goldenseal administration prior to the midazolam administration.
  Interventions: Drug: Midazolam Hcl 1Mg/Ml Inj; Dietary Supplement: Goldenseal (Hydrastis canadensis)

INTERVENTIONS:
Drug: Midazolam Hcl 1Mg/Ml Inj — 0.5 mL of an intravenous solution (1 mg/mL) will be administered.
  Other Names: Versed
Dietary Supplement: Goldenseal (Hydrastis canadensis) — Goldenseal (Solaray; Lot #1020199) is supplied as dried root powder in vegetable capsules, each containing 550 mg of herbal content. Goldenseal capsules will be administered with 240 mL of water.
  Arms: Study Arm 2: Acute Goldenseal Exposure; Study Arm 3: Chronic Goldenseal Exposure

SUMMARY:
Supplements containing goldenseal, a perennial herb native to North America, have consistently ranked among the top 20 highest selling natural products throughout the last decade. Goldenseal products are marketed as licensed natural health products in Canada and as dietary supplements in the United States. Natural products made from dried roots of the goldenseal plant are purported to have therapeutic value and are used to self-treat a range of medical complications, including the common cold, allergic rhinitis, and digestive disorders, such as diarrhea and constipation. Based on a previous clinical study, goldenseal have been shown to precipitate pharmacokinetic interactions with metformin in healthy volunteers. This follow-up study aims to evaluate the goldenseal-metformin interaction in type 2 diabetic patients. Results from this proposed clinical study will (1) characterize the pharmacokinetic interaction between the botanical dietary supplement goldenseal and anti-diabetic drug metformin, (2) provide evidence-based recommendations to mitigate drug interaction risks, and (3) contribute to the development of a comprehensive strategy for effectively assessing other potential natural-product drug interactions.

DETAILED DESCRIPTION:
Many patient groups, including those afflicted with cardiovascular disease, cancer, HIV/AIDS, hepatitis C, and diabetes, often supplement their prescribed pharmacotherapeutic regimens with herbal and other natural products, raising concern for adverse interactions. Unlike for drug-drug interactions, rigorous, harmonized guidelines for assessing the risk of natural product-drug interactions do not exist. The NCCIH-funded Center of Excellence for Natural Product Drug Interaction (NaPDI) Research was established in September 2015. The mission of the NaPDI Center is to provide leadership in the identification, evaluation, and dissemination of potential clinically meaningful pharmacokinetic natural product-drug interactions. Goldenseal is one of four high priority natural products selected by the NaPDI Center for further evaluation for drug interaction potential.

A recent clinical study completed by researchers at the NaPDI center showed that a well-characterized, adulterant- and contaminant-free goldenseal product administered to 16 healthy volunteers (3 g daily by mouth for 6 consecutive days) resulted in a significant decrease (23%) in metformin systemic exposure [area under the plasma concentration-time curve (AUC)] with no change in half-life or renal clearance. Based on these clinical observations, along with complementary in vitro data, the current working hypothesis is that goldenseal interacts with intestinal organic cation transporter 1 to alter metformin disposition. These observations may have clinical implications for diabetic patients, as metformin is the first-line treatment and most prescribed anti-diabetic medication for type 2 diabetes. The objective of this study is to assess the potential for goldenseal to alter the pharmacokinetics and clinical effects of standard metformin treatment in well-controlled adult type 2 diabetic patients.

Transporter inhibition represents an understudied mechanism of natural product-drug interactions. The proposed clinical study will be the first of its kind to evaluate whether such pharmacokinetic interactions can potentially affect clinical outcomes. The knowledge gained from these efforts will ultimately build upon a systematic framework for effectively studying other transporter-mediated natural product-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* are 18-65 years old and healthy
* have been medically diagnosed with Type 2 diabetes and currently taking metformin (1- 2 g daily), but otherwise healthy as determined by the study physician
* have an HbA1c < 8% as determined by laboratory analysis on initial screening
* are not taking any medications, dietary/herbal supplements, or citrus juices that can interfere with your ability to eliminate the study drugs and goldenseal from your body
* are willing to stop consuming alcohol, caffeinated beverages or other caffeine- containing products the evening before and the morning of the first day of each study arm
* are female and are willing to use an acceptable method of birth control that does not include oral birth control pills or patches (such as abstinence, copper IUD, condom)
* can provide written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

* have an HbA1c ≥ 8%
* have other chronic illnesses other than type 2 diabetes (e.g., type 1 diabetes, kidney disease, hepatic disease, uncontrolled hypertension, coronary artery disease, chronic obstructive pulmonary disease, cancer, or HIV/AIDS)
* have a hematologic (blood) disorder
* have a history of drug or alcohol abuse
* have any major psychiatric illness
* are pregnant or breastfeeding
* have a history of intolerance or allergy to midazolam or goldenseal products
* are taking concomitant medications, both prescription and non-prescription (including dietary supplements/herbal products) known to alter the pharmacokinetics of either study drug or goldenseal constituents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen JT, Tian DD, Tanna RS, Hadi DL, Bansal S, Calamia JC, Arian CM, Shireman LM, Molnar B, Horvath M, Kellogg JJ, Layton ME, White JR, Cech NB, Boyce RD, Unadkat JD, Thummel KE, Paine MF. Assessing Transporter-Mediated Natural Product-Drug Interactions Via In vitro-In Vivo Extrapolation: Clinical Evaluation With a Probe Cocktail. Clin Pharmacol Ther. 2021 May;109(5):1342-1352. doi: 10.1002/cpt.2107. Epub 2020 Dec 23. PMID 33174626
- [Background] Liang X, Giacomini KM. Transporters Involved in Metformin Pharmacokinetics and Treatment Response. J Pharm Sci. 2017 Sep;106(9):2245-2250. doi: 10.1016/j.xphs.2017.04.078. Epub 2017 May 8. PMID 28495567
- [Derived] Nguyen JT, Arian CM, Tanna RS, Cherel MG, Layton ME, White JR, Thummel KE, Paine MF. The Pharmacokinetic Interaction Between Metformin and the Natural Product Goldenseal Is Metformin Dose-Dependent: A Three-Arm Crossover Study in Adults With Type 2 Diabetes. Clin Transl Sci. 2025 Feb;18(2):e70120. doi: 10.1111/cts.70120. PMID 39943692

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A washout period of ≥7 days between each arm was implemented in the study design.
Groups:
- Midazolam Alone - Washout - Midazolam + Acute Goldenseal - Washout - Midazolam + Chronic Goldenseal: Twenty-two adults (12 males, 10 females) with type 2 diabetes participated in this three-arm, crossover study to assess a pharmacokinetic natural product-drug interaction. In arm 1 (midazolam alone), participants were administered a single dose of midazolam (0.5 mg) intravenously via a peripherally inserted catheter; at this time, participants were instructed to co-administer their entire daily dose of metformin orally. For Arm 2 (midazolam + acute goldenseal exposure), the same 22 participants were administered a single dose of goldenseal (3.3 g) orally 30 minutes prior to administration of midazolam and metformin. For Arm 3 (chronic goldenseal exposure), participants self-administered goldenseal (1.1 g) orally three times daily for 27 days. On the 28th day, participants were administered the goldenseal three times daily, as well as the single dose of midazolam and metformin. Plasma and urine were collected from 0-24 hours post-midazolam administration for all 3 arms of the study. A washout period of 7 days separated each arm to ensure appropriate washout of midazolam. Participants continued their routine administration of metformin as prescribed throughout the duration of the study without interruption in pharmacotherapy.
  Midazolam HCl 1mg/mL inj: 0.5 mL of intravenous solution
  Goldenseal (Hydrastis canadensis) 550 mg capsules: dried root powder in vegetable capsules (Solaray; Lot #1020199)
Period: Overall Study
Arm/Group | Midazolam Alone - Washout - Midazolam + Acute Goldenseal - Washout - Midazolam + Chronic Goldenseal
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Midazolam Alone - Washout - Midazolam + Acute Goldenseal - Washout - Midazolam + Chronic Goldenseal
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Metformin AUC
Description: Area under the plasma concentration time curve of metformin
Time Frame: Before and 20 minutes, 40 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, and 12 hours after midazolam administration.
Population: All 22 participants completed the 3 arms of the study (baseline, acute goldenseal exposure, and chronic goldenseal exposure).
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*hr/mL
Groups:
- Study Arm 1: Baseline: Twenty-two type 2 diabetic subjects (12 men, 10 women) were administered a single dose of midazolam (0.5 mg) intravenously via a peripherally inserted catheter in conjunction with their daily oral administration of metformin. Plasma and urine were collected from 0-24 hours post-midazolam administration. Participants self-administered their metformin as prescribed throughout the entirety of the study without interruption in pharmacotherapy.
  Midazolam HCl 1 mg/mL inj: 0.5 mL of an intravenous solution was administered.
- Study Arm 2: Acute Goldenseal Exposure: For Arm 2, the same 22 subjects were administered a single dose of goldenseal (3.3 g) orally 30 minutes prior to administration of midazolam and metformin. Plasma and urine were collected in a manner identical to that in Arm 1. With respect to midazolam administration, a washout period of 7 days separated Arm 2 from Arm 1.
  Midazolam HCl 1 mg/mL inj: 0.5 mL of an intravenous solution was administered.
  Goldenseal (Hydrastis canadensis): goldenseal (Solaray; Lot #1020199) was supplied as dried root powder in vegetable capsules, each containing 550 mg of herbal content. Goldenseal capsules were administered with 240 mL of water.
- Study Arm 3: Chronic Goldenseal Exposure: For Arm 3, the same 22 subjects self-administered goldenseal (1.1 g) orally three times daily for 27 days. On the 28th day, participants were administered the goldenseal three times daily, as well as the single dose of midazolam and metformin. Plasma and urine were collected in a manner identical to that in Arm 1 and 2. A designated washout period for midazolam was not necessary to separate Arm 3 since there will be 27 days of goldenseal administration prior to the midazolam administration.
  Midazolam HCl 1mg/mL inj: 0.5 mL of an intravenous solution was administered.
  Goldenseal (Hydrastis canadensis): Goldenseal (Solaray; Lot #1020199) was supplied as dried root powder in vegetable capsules, each containing 550 mg of herbal content. Goldenseal capsules were administered with 240 mL of water.
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
Number analyzed (Participants) | 22 | 22 | 22
mcg*hr/mL | 59.6 [52.0 to 68.5] | 54.5 [48.2 to 61.7] | 57.3 [50.3 to 65.3]
Statistical Analysis 1: Comparison: Study Arm 1: Baseline vs Study Arm 2: Acute Goldenseal Exposure vs Study Arm 3: Chronic Goldenseal Exposure; The predefined no effect range was 0.80-1.25; that is, if the geometric mean ratio lay outside this range, a pharmacokinetic interaction was evident; Test type: Other; AUC ratio (geometric mean) = 0.88, 90% CI 2-sided [0.82 to 0.96]

2. Primary Outcome: Metformin Cmax
Description: maximum concentration of metformin
Time Frame: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
Number analyzed (Participants) | 22 | 22 | 22
nM | 8.92 [7.86 to 10.1] | 8.36 [7.55 to 9.27] | 8.26 [7.37 to 9.25]
Statistical Analysis 1: Comparison: Study Arm 1: Baseline vs Study Arm 2: Acute Goldenseal Exposure vs Study Arm 3: Chronic Goldenseal Exposure; Test type: Other — The predefined no effect range was 0.80-1.25; that is, if the geometric mean ratio lay outside this range, a pharmacokinetic interaction was evident; Cmax ratio (geometric mean) = 0.93, 90% CI 2-sided [0.85 to 1.01]

3. Secondary Outcome: Metformin Half-Life
Description: half-life of metformin
Time Frame: 0-24h
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Groups:
- Study Arm 1: Baseline: Twenty type 2 diabetic subjects (10 men, 10 women) will be administered a single dose of midazolam (0.5 mg) intravenously via a peripherally inserted catheter in conjunction with their daily oral administration of metformin. Plasma and urine will be collected from 0-24 hours post-midazolam administration. Participants will take their metformin as prescribed for the entirety of the study with no interruption in pharmacotherapy.
  Midazolam Hcl 1Mg/Ml Inj: 0.5 mL of an intravenous solution (1 mg/mL) will be administered.
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
Number analyzed (Participants) | 22 | 22 | 22
hours | 4.73 [4.18 to 5.35] | 4.70 [4.22 to 5.23] | 4.79 [4.27 to 5.37]
Statistical Analysis 1: Comparison: Study Arm 1: Baseline vs Study Arm 2: Acute Goldenseal Exposure vs Study Arm 3: Chronic Goldenseal Exposure; Test type: Other; Half-life ratio (geometric mean) = 1.01, 90% CI 2-sided [0.93 to 1.07]

4. Secondary Outcome: Metformin Renal Clearance
Description: renal clearance of metformin
Time Frame: 0-24h
Measure: Geometric Mean (90% Confidence Interval); unit: mL / min
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
Number analyzed (Participants) | 22 | 22 | 22
mL / min | 259 [203 to 331] | 249 [200 to 309] | 250 [199 to 314]
Statistical Analysis 1: Comparison: Study Arm 1: Baseline vs Study Arm 2: Acute Goldenseal Exposure vs Study Arm 3: Chronic Goldenseal Exposure; Test type: Other; Renal clearance ratio (geometric mean) = 0.97, 90% CI 2-sided [0.84 to 1.12]

5. Secondary Outcome: Midazolam AUC
Description: area under the concentration vs. time curve of midazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*hr/mL
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
Number analyzed (Participants) | 22 | 22 | 22
mcg*hr/mL | 31.9 [27.1 to 37.7] | 31.1 [26.4 to 36.5] | 29.7 [25.7 to 34.3]
Statistical Analysis 1: Comparison: Study Arm 1: Baseline vs Study Arm 2: Acute Goldenseal Exposure vs Study Arm 3: Chronic Goldenseal Exposure; Test type: Other; AUC ratio (geometric mean) = 0.97, 90% CI 2-sided [0.81 to 1.15]

ADVERSE EVENTS:
Time Frame: All participants were monitored up to whenever they completed the final arm of the study, which was on average ~2 months.
Arm/Group | Study Arm 1: Baseline | Study Arm 2: Acute Goldenseal Exposure | Study Arm 3: Chronic Goldenseal Exposure
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 9/22 | 4/22 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Arm 1: Baseline (N=22) | Study Arm 2: Acute Goldenseal Exposure (N=22) | Study Arm 3: Chronic Goldenseal Exposure (N=22)
presyncope (Nervous system disorders) | 9 | 2 | 2
emesis (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT05081583/Prot_SAP_000.pdf